CLINICAL TRIAL: NCT04803318
Title: Trametinib Combined With Everolimus and Lenvatinib in the Treatment of Recurrent/Refractory Advanced Solid Tumors: a Phase II Clinical Trial
Brief Title: Trametinib Combined With Everolimus and Lenvatinib for Recurrent/Refractory Advanced Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZ3TKI-011
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor, Adult; Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma;Lung Cancer; Trametinib; Everolimus; Lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Everolimus; lenvatinib; Angiogenesis

STUDY DESIGN:
Intervention Model Description: To treat recurrent or refractory advanced solid tumors with multiple targeting drugs that inhibit several critical signaling pathways in cancer cells.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Combination treatment of 3 inhibitors (Experimental): Oral administration of 3 signaling pathways inhibitors: Mek inhibitor Trametinib, mTOR inhibitor Everolimus, and angiogenesis inhibitor Lenvatinib on refractory advanced solid tumors.
  Interventions: Drug: Combination of three inhibitors Trametinib, Everolimus and Lenvatinib

INTERVENTIONS:
Drug: Combination of three inhibitors Trametinib, Everolimus and Lenvatinib — Oral administration of three inhibitors including Trametinib, Everolimus and Lenvatinib.
  Other Names: Combination of 3 signaling pathway inhibitors specific to MEK, mTOR, and angiogenesis.

SUMMARY:
To study the clinical effect of Trametinib combined with Everolimus and Lenvatinib in the treatment of Recurrent/Refractory advanced solid tumors.

DETAILED DESCRIPTION:
The tumor diameter was measured and the efficacy was evaluated after treatment with Trametinib combined with Everolimus and Lenvatinib.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent/Refractory advanced solid tumors
* Age between 18 and 85 years
* Expected life expectancy is greater than three months

Exclusion Criteria:

* Benign tumor
* Life expectancy is less than three months
* Serious medical commodities
* others

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2037-01-01 (Estimated)

PRIMARY OUTCOMES:
Assessing Incidence of Treatment-Emergent Adverse Events during the treatment and various responses to the treatment. | up to 36 months

SECONDARY OUTCOMES:
Assessing progress free survival | 48 months
Assessing overall survival | 48 months
  Assessing overall time to survival.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided